CLINICAL TRIAL: NCT06271681
Title: Evaluation of PCV21 Vaccination Among PPSV23-experienced, Immunocompromised Elderly Veterans
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Sierra Nevada Health Care System (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Amneet Rai, Associate Chief of Pharmacy for Informatics, Education, Health Outcomes, and Research, VA Sierra Nevada Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2120135-1
Record Dates: First submitted 2024-01-04; First posted 2024-02-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Pneumococcal Vaccines; Immunosuppression
Keywords: immunosuppression; pneumococcal vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All participants (Other): This will be a single population open label trial evaluating immune response to PCV21 in subjects with immunocompromising conditions or receiving immunosuppressive medications.
  Interventions: Drug: 21-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Drug: 21-valent pneumococcal conjugate vaccine — FDA approved pneumococcal vaccines 21 valent conjugate vaccine administered at enrollment
  Other Names: PCV21

SUMMARY:
The investigators will evaluate the immune response of immunocompromised adults, who have previously received at least 1 dose of 23-valent pneumococcal polysaccharide vaccine, to the booster with of 21-valent pneumococcal conjugate vaccine . Immune response will be assessed by opsonophagocytic assay reactivity.

DETAILED DESCRIPTION:
Recommendations for optimal vaccination strategies in immunocompromised patients has been limited. Strategies focused on utilizing a conjugate vaccine alone, as either initial vaccination or booster dosing, have not demonstrated significant increased antibody expression in immunocompromised patients[7]. Strategies where immunocompromised patients were vaccinated with a conjugate vaccine followed by polysaccharide vaccine have demonstrated that 50% of individuals achieve functional antibodies[7]. Since improved antibody response in naive patients has been seen in combination vaccination, we aim to test this strategy for boosting in previously vaccinated immunocompromised patients. The 15 valent Pneumococcal Conjugate Vaccine (PCV15) is available for use in adults and contains S. Pneumoniae serotypes 1, 3, 4, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F and 33F [5].

In this study we postulate that booster dosing with PCV21 in immunocompromised adults who are at least 5 years from receipt of PPSV23 will elicit a strong immune response represented by change in serotype specific OPA GMT from baseline to 4 weeks post booster vaccine completion. We will specifically evaluate the change in pneumococcal opsonophagocytic activity at baseline to 6 months (Pn-OPA) for S. Pneumoniae serotypes 3, 6A, 15A, 19A, 20A, 23A, 31, 35B, 9n, 11A, and 22F. These specific serotypes have been selected due to current disease burden trends, to address current gaps in data, and have been identified as the most relevant for PCV development underway.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets the CDC definition of an immunocompromising condition

  o chronic renal failure, congenital or acquired asplenia, generalized malignancy, HIV infection, Hodgkin disease, iatrogenic immunosuppression, leukemia, lymphoma, multiple myeloma, nephrotic syndrome, sickle cell disease or other hemoglobinopathies, and solid organ transplant.
* Have received at least 1 dose of PPSV23

Exclusion Criteria:

* Less than 5 years since last receipt of PPSV23 validated to patient medical record and Immunize Nevada Website
* Previous administration of PCV20
* Previous administration of PCV13
* Previous administration of PCV15
* Less than 14 days since administration of any COVID19 vaccination
* Previous history of Invasive Pneumococcal Disease (IPD)
* Antibiotic treatment within the previous 90 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in opsonophagocytic assay (OPA) geometric mean titers (GMT) | 24 months
  Evaluation of the change fold increase in S. Pneumonia OPA GMT from baseline to 24 weeks after the administration of a pneumococcal vaccine booster series consisting of PCV15 followed by PPSV23 8 weeks later for S. Pneumoniae serotypes 1, 3, 4, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F and 33F

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not planned to be made available at this time.